CLINICAL TRIAL: NCT01274429
Title: Peanut Oral Immunotherapy (OIT) - Initial Pilot Study in Adults
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2314
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2017-03

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; Immunotherapy; OIT
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label peanut flour (Experimental): Orally ingested peanut flour administered in gradually increasing doses up to a maximum maintenance dose.
  Interventions: Drug: Peanut flour

INTERVENTIONS:
Drug: Peanut flour — Peanut flour that is ingested daily and administered in gradually increasing amounts up to a maximum maintenance dose.
  Other Names: Peanut OIT

SUMMARY:
The goal of this study is to produce a new treatment that would benefit adult subjects by lowering the risk of anaphylactic reactions (desensitization), and changing the peanut-specific immune response in subjects who have peanut allergy (tolerance). This project is designed to study the innovative idea that oral immunotherapy (OIT), the ingestion of small increasing amounts of food allergen, will desensitize subjects with peanut hypersensitivity by regulating their mucosal and systemic immune reactivity and cause long-term tolerance.

DETAILED DESCRIPTION:
The goal of this proposal is to produce a new treatment that would benefit subjects who have peanut allergy by lowering the risk of anaphylactic reactions (desensitization), and changing the peanut-specific immune response in subjects who have peanut allergy (tolerance). This is a research study to test stimulation of the immune system to improve peanut allergy. The approach the investigators will use for peanut allergy is called desensitization. A person becomes desensitized to a food by taking small, increasing amounts of the food to help the body become used to the food so that it no longer causes a severe allergic reaction.

The study also looks at the safety and immune system effects of the investigational study product, peanut protein. The word "investigational" means the study product is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA).

This project is designed to study if peanut oral immunotherapy (POIT) will desensitize subjects with peanut hypersensitivity by regulating their oral and systemic immune reactivity and cause long-term tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years of age of any gender, race, or ethnicity.
* Diagnosis of peanut allergy OR convincing clinical history of peanut allergy.
* Detectable serum peanut -specific Immune globin E(IgE) level (CAP-FEIA ≥ 0.35 kU/L) and a positive skin prick test (SPT) to peanut.
* Participant willing to use effective method of contraception if female for the duration of the study, not pregnant or lactating, and not planning to become pregnant.
* Positive reaction to ≤ 2 gm peanut protein on entry challenge.

Exclusion Criteria:

* History of severe anaphylaxis to peanut per current National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) allergic reaction toxicity grading.
* Known sensitivity or intolerance to Oats.
* FEV1 value <80% predicted or any clinical features of moderate or persistent asthma per 2007 National Heart Lung and Blood Institute (NHLBI) guidelines.
* Exacerbation of asthma in the past year requiring hospitalization or greater than 1 emergency department (ED) visit for asthma in the past 6 months.
* Use Beta-blockers, ACE inhibitors, angiotensin receptor blocker (ARB) , or calcium channel blockers, xolair, or immunological treatments.
* Uncontrolled hypertension per JNC 7 Guidelines (BP > 145/95 seated readings on each of two or more office visits).
* Active eosinophilic gastrointestinal disease which could be exacerbated by peanut oral immunotherapy.
* Chronic diseases such as diabetes, liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, blood disorders, or history of ischemic cardiovascular disease, or other conditions that in the opinion of the Investigator make the subject unsuitable for induction of food allergy reactions.
* Unable to speak English.
* Inability to discontinue antihistamines prior to food challenges and skin prick tests.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — Duke University
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Peanut Flour
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study closed do to lack of funding | 5

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Peanut Flour
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 19.5 [18.8 to 21.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Determine Whether This Peanut OIT Protocol Lowers Their Risk of Anaphylactic Reactions and Causes Long-term Tolerance.
Description: Assess mg of peanut tolerated on double-blind placebo-controlled food challenge as a measure of desensitization and tolerance
Time Frame: 2-3 years
Population: No subjects reached the end of study food challenge prior to closure of the study and therefore no data was collected towards this endpoint.
Arm/Group | Open Label Peanut Flour
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine the Effect That PNOIT Has on the Peanut-specific Cellular and Humoral Response in Peanut-allergic Subjects.
Description: Measure changes over the course of treatment in serum specific IgE and IgG4, skin prick tests, TH1 and TH2 cytokines, and CD4+ CD25+ FoxP3+ regulatory T cells
Time Frame: 2-3 years
Population: No subjects reached the end of study prior to closure of the study and therefore no end of treatment mechanistic data was collected in order to compare against the baseline.
Arm/Group | Open Label Peanut Flour
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Open Label Peanut Flour
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Peanut Flour (N=5)
Vomiting (Gastrointestinal disorders) | 0
Diarrhea (Gastrointestinal disorders) | 1
Erythematous rash (Skin and subcutaneous tissue disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0
Oropharyngeal itching (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0
Nose itch (Respiratory, thoracic and mediastinal disorders) | 1
Skin itch (Skin and subcutaneous tissue disorders) | 0
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 0
Eye itch (Eye disorders) | 0
Eye tearing (Eye disorders) | 0
Hives (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination due to lack of funding prior to any subjects reaching the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No